CLINICAL TRIAL: NCT04055220
Title: A Randomized, Placebo-controlled, Double-blinded, Multicentre Study Evaluating the Efficacy and Safety of Regorafenib as Maintenance Therapy After First-line Treatment in Patients With Bone Sarcomas
Brief Title: Efficacy and Safety of Regorafenib as Maintenance Therapy After First-line Treatment in Patients With Bone Sarcomas
Acronym: REGOSTA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Leon Berard (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REGOSTA (ET18-272)
Record Dates: First submitted 2019-08-05; First posted 2019-08-13 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Bone Sarcoma; Osteosarcoma; Ewing Sarcoma; Chondrosarcoma; Undifferentiated Pleomorphic Sarcoma; Leiomyosarcoma; Angiosarcoma
Keywords: Maintenance therapy; First line therapy; Regorafenib; Randomization; Double-blinded; Placebo controlled; Relapse-free survival; Time to treatment failure; Overall survival; Quality of life; Compliance; Bone sarcoma; Osteosarcoma; Efficacy; Complete response; Tyrosine kinase inhibitor; Multi-target inhibitor; Safety
MeSH Terms: conditions — Bone Neoplasms; Osteosarcoma; Sarcoma, Ewing; Chondrosarcoma; Histiocytoma, Malignant Fibrous; Leiomyosarcoma; Hemangiosarcoma; Patient Compliance; Pathologic Complete Response | interventions — regorafenib; Standard of Care

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Regorafenib (Experimental): Treatment will be divided in 28 days cycles, including a 21-day period of treatment by regorafenib followed by a 7-day period of rest.
  In case of toxicity, dose can be reduced or treatment interrupted according to Specific Product Characteristics (SPC).
  Patients can receive up to a maximum of 13 cycles (maximum treatment period : 12 Months).
  Interventions: Drug: Treatment by Regorafenib
- Placebo (Placebo Comparator): Treatment will be divided in 28 days cycles, including a 21-day period of treatment by placebo followed by a 7-day period of rest.
  In case of toxicity, dose can be reduced or treatment interrupted according to Specific Product Characteristics (SPC).
  Patients can receive up to a maximum of 13 cycles (maximum treatment period : 12 Months).
  Interventions: Drug: Treatment by Placebo

INTERVENTIONS:
Drug: Treatment by Regorafenib — Treatment for 13 cycles (12 months) maximum.
  During each cycle, patient will take once a day, during 21 days, followed by 7 days without treatment :
  * 3 tablets daily, corresponding to a total of 120 mg of Regorafenib (3 weeks out of 4 weeks) in patients ≥ 16 years old and patients < 16 years old with BSA ≥ 1.70m²;
  * 2 tablets daily corresponding to a total of 80 mg of Regorafenib (3 weeks out of 4 weeks) in patients < 16 years old with 1.30m² ≤ BSA < 1.70m²;
  Other Names: Stivarga
  Arms: Regorafenib
Drug: Treatment by Placebo — Treatment for 13 cycles (12 months) maximum.
  During each cycle, patient will take once a day, during 21 days, followed by 7 days without placebo treatment :
  * 3 placebo tablets (3 weeks out of 4 weeks) in patients ≥ 16 years old and patients < 16 years old with BSA ≥ 1.70m²;
  * 2 placebo tablets (3 weeks out of 4 weeks) in patients < 16 years old with 1.30m² ≤ BSA < 1.70m²;
  Other Names: Standard of care
  Arms: Placebo

SUMMARY:
This is a randomized, double-blinded, 2 arms study concerning patients with bone sarcoma after the first line therapy.

In the first arm, patients will be treated with regorafenib for a maximum of 12 months as maintenance therapy after first line therapy, whereas in the second arm, patients will be treated with placebo (standard of care).

The comparison between this two arms will allow to determine whether or not regorafenib is efficient for disease control, in terms of Relapse-Free Survival improvement.

DETAILED DESCRIPTION:
Bone sarcomas are rare primary bone cancers, although, their frequency has been increasing by 0.3% per year over the last decade. They include a very large number of tumour types belonging to the family of primary malignant bone tumours and originate from bone as Osteosarcomas (OS), Chondrosarcomas (CS), Fibrosarcomas, Chordomas, …

Current conventional treatments for OS combine chemotherapy and surgery. Chemotherapy treatment is commonly given for OS over a period of 6-10 months, with a period of preoperative chemotherapy, to facilitate local surgical treatment. The conventional cocktail used in OS is composed by a minimum of three drugs (reference combination: methotrexate, doxorubicin and cisplatin (MAP)).

The currently recommended treatments for Ewing sarcomas (for both localized and metastatic diseases) consist of multimodal approaches including surgery and/or radiotherapy associated to neoadjuvant and adjuvant chemotherapy, comprising respectively from 3 to 6, and then from 6 to 10 cycles. Doxorubicin, cyclophosphamide, ifosfamide, vincristine, dactinomycin and etoposide are considered as the most active substances. Current trials require combination chemotherapies, and most of them are based on the combination of 5-6 of these substances.

Concerning chondrosarcomas, the treatment is adapted according to the subtype. Thus, the treatment regimen for mesenchymal chondrosarcomas and dedifferentiated chondrosarcomas differs. Indeed, an Ewing-type chemotherapy regimen is usually suggested to treat mesenchymal chondrosarcomas while dedifferentiated chondrosarcomas are often treated as high-grade bone sarcoma, with systemic and local therapies.

Compared with surgery alone, multimodal treatment of high-grade sarcomas increases disease-free survival probabilities from only 10%-20% to 50-65% depending on the bone sarcoma type. In general, despite second-line treatment, the prognosis of recurrent disease has remained poor, with long-term post-relapse survival of <20%.

The outcome of bone sarcoma has been dramatically improved by the addition of chemotherapy in the 70' and 80' but has remained remarkably stable in the last 3 decades, with a survival rate largely plateaued, despite introduction of novel regimens, both in localized and metastatic disease, in children and in adults. Primary bone cancer presented challenges in new drug development partly because of their rarity and heterogeneity. Thus, improving treatments for these diseases is a high priority, but advances have been few in recent years. In this context, maintenance therapy may be an interesting option as a way to prolong the benefit of first-line chemotherapy.

Regorafenib may play a role in the maintenance setting for bone sarcomas (as improved Progression-Free Survival and sustained responses were observed in the REGOBONE study) in maintaining the initial response to standard treatments and delaying the need for further treatment at relapse, while exerting a manageable associated toxicity and minimal negative impact on health-related quality of life.

Currently there is no available agent used as maintenance therapy after first-line treatments. In the context of a clinical trial with close monitoring, it is, thus, acceptable to consider a placebo-control group.

On this basis, this study propose to conduct a double-blinded randomized controlled trial to evaluate the efficacy of regorafenib versus placebo in the treatment of patients with bone sarcomas, who have no evidence of disease after standard multimodal treatments based on the histological subtype.

The main goal of the present study is then to explore whether sequential addition of regorafenib after completion of a standard treatment in patients with bone sarcomas would improve outcomes in term of event-free-survival (EFS) defined by local or distant recurrence of the disease.

Results will be stratified on the "high-risk" versus "low-risk" of relapse. As response to neoadjuvant chemotherapy and metastatic status at time of diagnosis are known to be important on patient's outcome, stratification will rely on a combined criteria taking into account these two factors. Thus, "high-risk" of relapse will be defined by the group of patients who are poor responders to neoadjuvant chemotherapy and/or in metastatic setting at diagnosis, whereas "low-risk" of relapse will be defined by the group of patients who have no metastatic disease at time of diagnosis and are good responders to neoadjuvant chemotherapy.

ELIGIBILITY:
INCLUSION CRITERIA :

I1. Age ≥ 12 years at the day of consenting to the study;

I2. Patients must have histologically confirmed diagnosis of primary bone sarcoma including but not limited to: Osteosarcomas, Ewing sarcomas, Chondrosarcomas, Undifferentiated Pleomorphic Sarcomas (UPS), Leiomyosarcomas (LMS) and Angiosarcomas;

I3. Prior treatment for localized or metastatic disease for bone sarcoma must have been completed, consisting of a standard multimodal treatment based on the histological subtype:

For OS, (excepted head and neck localisations), neoadjuvant and/or adjuvant chemotherapy should include methotrexate-based regimen for patients < 18 years old; patients ≥ 18 years old may have received either methotrexate-based regimen or anthracycline and cisplatin-based regimen For head and neck OS, neoadjuvant and/or adjuvant chemotherapy should include adriamycin, cisplatin or ifosfamide-based regimen.

For non-OS, neoadjuvant and/or adjuvant chemotherapy should include adriamycin and/or cisplatin-based regimen.

I4. Recovery to NCI-CTCAE v5 Grade 0 or 1 level or recovery to baseline preceding the prior treatment from any previous drug/procedure related toxicity (except alopecia, anaemia, and hypothyroidism);

I5. Interval between the last chemotherapy administration and the date of randomisation: at least 4 weeks but no longer than 2 months;

I6. Confirmed complete remission or no evidence of disease (for metastatic disease);

Patients with pulmonary micro nodules can be included provided they do not meet the following criteria:

* At least one lung nodule of 10mm or more
* And/or at least two nodules well limited between 6-9mm
* And/or at least 5 nodules well limited of 5mm or less All the other situations will be considered as doubtful lesions except in case of metastatic disease confirmed during the lung surgery of the residual lung lesions after pre-operative chemotherapy. If no other metastatic localisation is detected at the initial staging, the patient will be considered as localised disease and eligible for randomisation.

I7. Life expectancy of greater than 12 months;

I8. Karnofsky Performance status ≥70 (patients younger than 18-year old) or ECOG performance status < 2 (adult patients) ;

I9. Patients must have adequate bone marrow, renal, and hepatic function, as evidenced by the following within 7 days of study treatment initiation:

* Absolute neutrophil count ≥ 1.5 Giga/l
* Platelets ≥ 100 Giga/l
* Haemoglobin≥ 9 g/dl
* Serum creatinine ≤ 1.5 x ULN
* Glomerular filtration rate (GFR) ≥30 ml/min/1.73m2 according to the Modified Diet in Renal Disease (MDRD) abbreviated formula
* AST and ALT ≤2.5 x ULN ( ≤5.0 × ULN for patients with liver involvement of their cancer)
* Bilirubin ≤1.5 X ULN
* Alkaline phosphatase ≤2.5 x ULN (≤5 x ULN in patient with liver involvement of their cancer). If Alkaline phosphatase > 2.5 ULN, hepatic isoenzymes 5-nucleotidase or GGT tests must be performed; hepatic isoenzymes 5-nucleotidase must be within the normal range and/or GGT < 1.5 x ULN.
* Lipase ≤1.5 x ULN
* Spot urine must not show ≥ 1 "+"protein in urine or the patient will require a repeat urine analysis. If repeat urinalysis shows 1 "+" protein or more, a 24-hour urine collection will be required and must show total protein excretion <1000 mg/24 hours

I10. INR/PTT ≤1.5 x ULN; Patients who are therapeutically treated with an agent such as warfarin or heparin will be allowed to participate provided that no prior evidence of underlying abnormality in coagulation parameters exists. Close monitoring of at least weekly evaluations will be performed until INR/PTT is stable based on a measurement that is pre-dose as defined by the local standard of care;

I11. Women of childbearing potential and male patients must agree to use adequate contraception (Appendix 4) for the duration of treatment and for 7 months (210 days) in WOCBP or 4 months (120 days) in men sexually active with WOCBP after the last dose of regorafenib;

I12. Women of childbearing potential must have a negative serum β-HCG pregnancy test within 7 days prior randomization and/or urine pregnancy test within 48 hours before the first administration of the study treatment;

I13. Patients, and their parents when applicable, must sign and date an informed consent document indicating that they have been informed of all the pertinent aspects of the trial prior to enrolment;

I14. Patients must be willing and able to comply with scheduled visits, treatment plan, laboratory tests and other study procedures;

I15. Patients covered by a medical insurance.

I16. Body Surface Area (BSA) ≥ 1.30m² at the time of consenting to the study.

NON-INCLUSION CRITERIA :

E1. Prior treatment with any VEGFR inhibitor (thus, any prior exposure to sunitinib, sorafenib, pazopanib, bevacizumab, or other VEGFR inhibitor);

E2. All soft tissue sarcomas (including but not limited to soft tissue osteosarcomas and Ewing soft tissue sarcomas) and chordomas;

E3. Prior history of other malignancies other than study disease (except for basal cell or squamous cell carcinoma of the skin or carcinoma in situ of the cervix) within 3 years prior to randomization;

E4. Cardiovascular dysfunction:

* Left ventricular ejection fraction (LVEF) < 50%,
* Congestive heart failure ≥ New York Heart Association (NYHA) class 2,
* Myocardial infarction < 6 months prior to first study drug administration,
* Cardiac arrhythmias requiring therapy (beta blockers or digoxin are permitted),
* Unstable (angina symptoms at rest) or new-onset angina within the last 3 months prior to first study drug administration;

E5. Uncontrolled hypertension (systolic blood pressure > 150mmHg or diastolic pressure > 90 mmHg despite optimal treatment);

E6. Arterial or venous thrombotic or embolic events such as cerebrovascular accident (including transient ischemic attacks), deep vein thrombosis, or pulmonary embolism within the last 6 months before the first study drug administration;

E7. Major surgical procedure, open biopsy or significant traumatic injury within 28 days before the first study drug administration;

E8. Ongoing infection > Grade 2 according to NCI-CTCAE v5;

E9. Known history of human immunodeficiency virus (HIV) infection;

Nota Bene: Subjects with diagnosed human immunodeficiency virus (HIV) are eligible to participate in the study if they meet the following criteria:

1. No history of acquired immunodeficiency syndrome (AIDS)-defining opportunistic infection within the past 12 months prior to enrolment;
2. No history of AIDS-defining cancers (e.g. Kaposi's sarcoma, aggressive B-cell lymphoma and invasive cervical cancer);
3. Subjects should be on established anti-retroviral therapy for at least 4 weeks and have an HIV viral load of < 400 copies/mL prior to enrolment;

E10. Active hepatitis B or C or chronic hepatitis B or C requiring treatment with antiviral therapy; Nota Bene: Subjects with a history of hepatitis B or C who have normal alanine aminotransferase (ALT) and are hepatitis B surface antigen negative and/or have undetectable HCV RNA are eligible;

E11. Dehydration according to NCI-CTC v5 Grade >1;

E12. Difficulties to swallow oral medication and/or any mal-absorption condition and/or any Gastrointestinal (GI) disease that may significantly alter the absorption of regorafenib (e.g., ulcerative diseases, uncontrolled nausea, vomiting, diarrhoea, malabsorption syndrome, or small bowel resection);

E13. Patients with seizure disorder requiring medication;

E14. Concurrent enrolment in another clinical trial in which investigational therapies are administered;

E15. Known hypersensitivity to the active substance or to any of the excipients;

E16. Pregnant women, women who are likely to become pregnant or are breast-feeding

E17. Patients with any psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule; those conditions should be discussed with the patient before registration in the trial;

E18. Patients with history of non-compliance to medical regimens or unwilling or unable to comply with the protocol;

E19. Interstitial lung disease with ongoing signs and symptoms at the time of informed consent;

E20. Non-healing wound, non-healing ulcer, or non-healing bone fracture;

E21. Patients with evidence or history of any bleeding diathesis, irrespective of severity;

E22. Any haemorrhage or bleeding event ≥ CTCAE v5 Grade 3 within 4 weeks prior to the first study drug administration;

E23. Clinically significant unrelated systemic illness (e.g., serious infection or significant cardiac, pulmonary, hepatic, or other organ dysfunction) that would compromise the patient's ability to tolerate study treatment or would likely interfere with study procedures or results;

E24. Patients using prohibited concomitant and/or concurrent medications (see section "Prohibited concomitant/concurrent treatments);

E25.Patients under tutorship or curatorship.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 168 (Estimated)
Dates: Start 2020-03-03 (Actual); Primary Completion 2026-10-01 (Estimated); Study Completion 2026-10-01 (Estimated)

PRIMARY OUTCOMES:
Relapse-Free Survival (RFS) | Up to 5 years
  RFS will be defined as the time from randomization to relapse, or death from any cause, whichever occurs first. Patients alive without relapse at the time of the analysis will be censored at the date of last tumour assessment. The Kaplan-Meier approach will be used to estimate median RFS for each study arm. The two-sided log-rank test, stratified on randomization stratification factors, will be used to compare RFS between the investigational arm and the control arm. The stratified Cox-regression (with proportional hazards) will be used to estimate the hazard ratio and to calculate the 95% confidence intervals of the hazard ratio.

SECONDARY OUTCOMES:
Time to Treatment Failure (TTF) | Up to 1 year
  TTF will be defined as the time from the date of randomization to the date of permanent discontinuation of the study treatment, whichever is the cause. Patient not known to have withdrawn treatment before 12 months (study treatment duration) will be censored at the time of treatment stop. TTF survival will be estimated using the Kaplan-Meier method, and will be described in terms of medians along with the associated 2-sided 95% confidence interval for the estimates.
Overall Survival (OS) | Up to 5 years
  OS will be defined as the time from date of randomization to the date of death, from any cause. Patient not known to have died at the time of analysis will be censored based on the last recorded date on which the patient was known to be alive. OS survival will be estimated using the Kaplan-Meier method, and will be described in terms of medians along with the associated 2-sided 95% confidence interval for the estimates.
Patient's Quality of Life (QoL) | Up to 5 years
  The patient's Quality of Life will be assessed using the EORTC QLQ-C30. Scores will be calculated at each time point according to the scoring manuals. Descriptive statistics will be used to evaluate baseline scores and evolution of scores from baseline to each time point (Every 3 months since baseline, then every 4 months after second year surveillance). Data will be compared between arms using the Student's t-test. The QoL data will also be presented graphically if deemed relevant.
Safety profile | Up to 5 years
  The safety will be described mainly on the frequency of adverse events coded using the common toxicity criteria (NCI-CTCAE v5.0) grade. Descriptive statistics will be provided for characterizing and assessing patient tolerance to treatment. Adverse events will be coded according to the MedDRA®.
Compliance To Treatment | Up to 1 year
  The compliance to treatment will be described using the proportion of patients requiring dose reduction and temporary or permanent treatment discontinuation.

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Yves BLAY, Principal Investigator — Centre Léon Bérard, Lyon; Florence DUFFAUD, Principal Investigator — Hôpital de la Timone (MARSEILLE); Sophie PIPERNO-NEUMANN, Principal Investigator — Institut Curie Paris
Locations (16):
- France (16):
  - Hôpital Jean Minjoz, Besançon
  - Institut Bergonié, Bordeaux
  - Centre Oscar Lambret, Lille
  - Centre Léon Bérard, Lyon
  - APHM - Hôpital Timone, Marseille
  - ICM Val d'Aurelle, Montpellier
  - Institut Curie, Paris
  - APHP Hôpital Cochin, Paris
  - Centre Hospitalier Universitaire de Poitiers, Poitiers
  - Centre Hospitalier Universitaire de Saint-Etienne (CHUSE), Saint-Etienne
  - ICO René Gauducheau, Saint-Herblain
  - Institut de Cancérologie Strasbourg Europe, Strasbourg
  - Centre Hospitalier Régional de Strasbourg Hautepierre, Strasbourg
  - IUCT-Oncopole, Toulouse
  - ICL Alexis Vautrin, Vandœuvre-lès-Nancy
  - Institut Gustave Roussy, Villejuif